CLINICAL TRIAL: NCT04860583
Title: Nephrocalcinosis in Very Low Birth Weight Infants: an Observational Study
Brief Title: Nephrocalcinosis in Very Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2021_001
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Infant; Premature, Light-For-Dates
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Renal ultrasound

SUMMARY:
Extremely premature children benefit from specific follow-up that requires high nutritional intake and the use of specific therapies that expose them to the risk of nephrocalcinosis. Other identified risk factors are extreme prematurity and intrauterine growth restriction.

The incidence of nephrocalcinosis in very premature infants is unclear, ranging from 7 to 64%. Most studies are observational and only few case-control studies can properly analyse the risk factors for nephrocalcinosis in significant populations that include only preterm infants.

This nephrocalcinosis of prematurity regresses spontaneously in more than half of the cases, but has been associated with a risk of long-term complications: impaired renal function, high blood pressure, etc. This is an aggravating factor in the context of prematurity, which has been associated with an increased risk of renal impairment and hypertension in childhood and adulthood.

For all these reasons, nutritional intakes and therapeutics are monitored very closely and a renal ultrasound is routinely performed at discharge at 35 weeks of corrected gestational age in all children who are born at a gestational age ≤ 32 weeks and/or birth weight ≤ 1500 g.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with a gestational age <= 32 weeks and/or birthweight <=1500g

Exclusion Criteria:

* Newborns with kidney malformation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born at the Croix-Rousse Hospital, Lyon, France between 01/01/2012 and 31/12/2017 with a gestational age <= 32 weeks and/or a birthweight <=1500g. Infants with a diagnosed kidney malformation are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of nephrocalcinosis | At week 35 of corrected gestational age
  Presence/absence of nephrocalcinosis will be checked by ultrasound

IPD SHARING:
Plan to Share IPD: Undecided